CLINICAL TRIAL: NCT03357796
Title: A Randomized, Open-label, Cross-over, 2-period Study to Assess the Relative Bioavailability Between 80 mg LY03005 Versus 50 mg Desvenlafaxine Comparator (Pristiq®) Under Fasting Condition After Single Dose Administration in Healthy Subjects
Brief Title: Relative Bioavailability (RBA) Study of LY03005 vs Pristiq®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY03005/CT-USA-104
Record Dates: First submitted 2017-11-21; First posted 2017-11-30 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-11

CONDITIONS: Major Depressive Disorder
Keywords: Depressive Disorder, Major; Depressive Disorder; Mood Disorders; Mental Disorders; Desvenlafaxine Succinate; Serotonin and Noradrenaline Reuptake Inhibitors; Neurotransmitter Uptake Inhibitors; Membrane Transport Modulators; Molecular Mechanisms of Pharmacological Action; Neurotransmitter Agents; Physiological Effects of Drugs; Antidepressive Agents; Psychotropic Drugs
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Mood Disorders; Mental Disorders | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: LY03005 cross-over to Pristiq® (Experimental): Subjects in Group A will receive an 80 mg oral dose of LY03005 and the subjects will stay in the CRU for 4 days (Period 1). After a washout period of up to 4 days, the subjects will be switched and will receive a 50 mg oral dose of desvenlafaxine (Pristiq®) comparator followed by a 4-day stay in the CRU (Period 2).
  Interventions: Drug: LY03005; Drug: Pristiq
- Group B: Pristiq® cross-over to LY03005 (Experimental): Subjects in Group B will receive a 50 mg oral dose of desvenlafaxine (Pristiq®) comparator and the subjects will stay in the CRU for 4 days (Period 1). After a washout period of up to 4 days, the subjects will be switched and will receive an 80 mg oral dose of LY03005 followed by a 4-day stay in the CRU (Period 2).
  Interventions: Drug: LY03005; Drug: Pristiq

INTERVENTIONS:
Drug: LY03005 — 80 mg, oral tablets, single dose
Drug: Pristiq — 50 mg, oral tablets, single dose
  Other Names: Desvenlafaxine

SUMMARY:
The objective of this study is to evaluate relative bioavailability between 80 mg LY03005 oral tablets and 50 mg Pristiq® oral tablets after a single dose of each drug in a cross-over 2-period design under fasting condition in healthy subjects between 18 and 50 years of age.

DETAILED DESCRIPTION:
Twenty (20) eligible subjects will be enrolled and assigned to either Group A or Group B at a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent and complying with study procedures;
2. Male and female subjects between the ages of 18 and 50 years;
3. Considered healthy as assessed by the principal investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs;
4. Nonsmoker, defined as not having smoked or used any form of tobacco in more than 6 months before Screening based on subject report;
5. Body mass index (BMI) of 19 to 28 kg/m2 inclusive and body weight not less than 50 kg;
6. Willing and able to adhere to study procedures and to be confined at the clinical research center.
7. All female subjects no matter of age must have a negative serum pregnancy test result at Screening. In addition, female subjects must meet one of the following 3 conditions: (i) postmenopausal for at least 2 years, (ii) surgically sterile based on subject report, or (iii) if child-bearing potential, practicing or agree to practice an effective method of birth control by using an acceptable method of contraception. Acceptable methods of birth control include intrauterine device (IUD), or double-barrier method (e.g., condom, diaphragm or cervical cap with spermicidal foam, cream, gel or suppository). Acceptable methods of birth control must be used for at least 14 days prior to the use of study drug during the study and within 1 month after the end of the study.

Exclusion Criteria:

1. Clinically significant past medical history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, ophthalmological, or drug hypersensitivity or any condition that in the judgement of the investigator will affect the study results or the subject's safety;
2. History of suicide attempt in the past 12 months and/or seen by the investigators as having a significant history of risk of suicide or homicide;
3. History or presence of malignancy other than adequately treated and cured basal cell skin cancer;
4. Clinically relevant illness within 1 month prior to the Screening Visit or at Screening Visit that may interfere with the conduct of this study;
5. Subjects with a mean systolic blood pressure >140 mmHg or a mean diastolic blood pressure of >90 mmHg at Screening after 3 measurements (after 5 minutes of rest in a sitting position);
6. Positive blood Screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
7. A history of seizure. However, a history of febrile seizure is allowed;
8. A hospital admission or major surgery within 30 days prior to Screening;
9. Participation in any other investigational drug trial within 30 days prior to Screening;
10. A history of prescription drug abuse or illicit drug use within 6 months prior to Screening;
11. A history of alcohol abuse according to medical history within 6 months prior to Screening;
12. A positive screen for alcohol and drugs of abuse;
13. Subjects with hypersensitivity to ODV or medicines containing ODV or its precursor venlafaxine;
14. Subjects who have participated in a previous clinical study of either LY03005 or ODV or medicines containing ODV or its precursor, venlafaxine within 30 days prior to Screening;
15. Unwillingness or inability to comply with food and beverage restrictions during study participation;
16. Donation of blood of more than 1 unit (approximate 450 mL) or blood products or acute loss of blood during the 90 days prior to Screening;
17. Use of prescription or over-the-counter (OTC) medications, and herbals (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at <3g/day is permitted until 24 hours prior to dosing).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) Assessment | PK Samples drawn at 0, 1,2,3,4, 6,8,10,12,24,32,48 and 72 hours after dosing in both Period 1 and Period 2.
  Area under the concentration-time curve (AUC) for the Pharmacokinetics (PK) of O-desmethyl-venlafaxine (ODV) from LY03005 and ODV from Pristiq will be determined.
Maximum concentration (Cmax) Assessment | PK Samples drawn at 0, 1,2,3,4, 6,8,10,12,24,32,48 and 72 hours after dosing in both Period 1 and Period 2.
  Maximum concentration (Cmax) for the Pharmacokinetics (PK) of O-desmethyl-venlafaxine (ODV) from LY03005 and ODV from Pristiq will be determined.

SECONDARY OUTCOMES:
Adverse Events Assessment | up to 35 days
  Collection of adverse events throughout the study as a measure of safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Sun, MD, PhD, MBA, Study Chair — Luye Pharma Group Ltd.
Locations (1):
- Clinilabs, Inc., Eatontown, New Jersey, United States

REFERENCES:
- See also: Drug Information — https://druginfo.nlm.nih.gov/drugportal/
- See also: Desvenlafaxine — https://druginfo.nlm.nih.gov/drugportal/name/Desvenlafaxine
- See also: Desvenlafaxine Succinate — https://druginfo.nlm.nih.gov/drugportal/name/desvenlafaxine%20succinate
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: Pristiq (Desvenlafaxine) Label - FDA — https://www.accessdata.fda.gov/drugsatfda_docs/label/2012/021992s030lbl.pdf